CLINICAL TRIAL: NCT03682705
Title: Rheumatoid Arthritis: A Phase 2 Study to Investigate the Safety and Efficacy of ABBV-105 Given Alone or in Combination With Upadacitinib (ABBV-599 Combination) With a Background of Conventional Synthetic DMARDs in Subjects With Active Rheumatoid Arthritis With Inadequate Response or Intolerance to Biologic DMARDs
Brief Title: A Study to Investigate the Safety and Efficacy of ABBV-105 Alone or in Combination With Upadacitinib (ABBV-599 Combination) in Participants With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-063; 2018-000666-10 (EudraCT Number)
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Elsubrutinib; ABBV-105; Upadacitinib; ABBV-599; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- ELS placebo/UPA placebo (Placebo Comparator): Placebo capsule for elsubrutinib once a day by mouth for 12 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 12 weeks
  Interventions: Drug: Placebo for elsubrutinib; Drug: Placebo for upadacitinib
- UPA 15 mg/ELS 60 mg (Experimental): 15 mg film-coated upadacitinib tablet once a day by mouth for 12 weeks; 60 mg elsubrutinib capsule once a day by mouth for 12 weeks
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- ELS 60 mg/UPA placebo (Experimental): 60 mg elsubrutinib capsule once a day by mouth for 12 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 12 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- ELS 20 mg/UPA placebo (Experimental): 20 mg elsubrutinib capsule once a day by mouth for 12 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 12 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- ELS 5 mg/UPA placebo (Experimental): 5 mg elsubrutinib capsule once a day by mouth for 12 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for 12 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib
- UPA 15 mg/ELS placebo (Experimental): 15 mg film-coated upadacitinib tablet once a day by mouth for 12 weeks; placebo capsule for elsubrutinib once a day by mouth for 12 weeks
  Interventions: Drug: Upadacitinib; Drug: Placebo for elsubrutinib

INTERVENTIONS:
Drug: Elsubrutinib — Elsubrutinib capsule will be administered orally.
  Other Names: ABBV-105
  Arms: ELS 20 mg/UPA placebo; ELS 5 mg/UPA placebo; ELS 60 mg/UPA placebo; UPA 15 mg/ELS 60 mg
Drug: Upadacitinib — Upadacitinib tablet will be administered orally.
  Other Names: ABT-494
  Arms: UPA 15 mg/ELS 60 mg; UPA 15 mg/ELS placebo
Drug: Placebo for elsubrutinib — Placebo capsule for elsubrutinib will be administered orally.
  Arms: ELS placebo/UPA placebo; UPA 15 mg/ELS placebo
Drug: Placebo for upadacitinib — Placebo tablet for upadacitinib will be administered orally.
  Arms: ELS 20 mg/UPA placebo; ELS 5 mg/UPA placebo; ELS 60 mg/UPA placebo; ELS placebo/UPA placebo

SUMMARY:
This was a phase 2 study to evaluate the safety and efficacy of elsubrutinib (ELS) and ABBV-599 (ELS plus upadacitinib [UPA]) vs placebo on a background of conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) for the treatment of signs and symptoms of rheumatoid arthritis (RA) at 12 weeks in biological disease-modifying anti-rheumatic drugs (bDMARD)-inadequate response (bDMARD-IR) or bDMARD-intolerant participants with moderately to severely active RA and to define optimal dose for further development.

DETAILED DESCRIPTION:
This was a 12-week, randomized, double-blind, parallel-group, Phase 2, dose exploratory, multicenter study. Participants who met eligibility criteria were randomized in a 3:2:2:2:2:1 ratio to 1 of 6 treatment groups: ABBV-599 [UPA 15 mg/ELS 60 mg]); ELS 60 mg/UPA placebo; ELS 20 mg/UPA placebo; ELS 5 mg/UPA placebo; UPA 15 mg/ELS placebo; and ELS placebo/UPA placebo. The study included a 35-day maximum screening period and a 12-week treatment period with 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for ≥ 3 months based on the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria for RA
* Participant meets the following minimum disease activity criteria:

  * ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits
  * High-sensitivity C-reactive protein (hsCRP) ≥ 3 mg/L (central lab) at Screening Visit
* Participants must have been treated for ≥ 3 months with ≥ 1 biologic disease-modifying anti-rheumatic drug (bDMARD) therapy but continue to exhibit active RA or had to discontinue due to intolerability or toxicity, irrespective of treatment duration
* Participants must have been receiving conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug
* Participants must have discontinued all bDMARDs prior to the first dose of study drug

Exclusion Criteria:

- Participant has prior exposure to any Janus Kinase (JAK) inhibitor for greater than 2 weeks (including but not limited to upadacitinib, tofacitinib, baricitinib, and filgotinib). A washout period of ≥ 30 days is required for any JAK inhibitor prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (115):
- United States (78):
  - Rheum Assoc of North Alabama /ID# 167382, Huntsville, Alabama
  - AZ Arthritis & Rheum Research /ID# 167446, Mesa, Arizona
  - SunValley Arthritis Center, Lt /ID# 213073, Peoria, Arizona
  - AZ Arthritis and Rheum Researc /ID# 167448, Phoenix, Arizona
  - St. Joseph Heritage Healthcare /ID# 167379, Fullerton, California
  - Purushotham, Akther & Roshan K /ID# 168121, La Mesa, California
  - Valerius Medical Group /ID# 168123, Los Alamitos, California
  - Sierra Rheumatology /ID# 167976, Roseville, California
  - Rheumatology Center of San Diego /ID# 170690, San Diego, California
  - Iraj Sabahi Research, Inc /ID# 201923, Turlock, California
  - Inland Rheum Clin Trials Inc. /ID# 167459, Upland, California
  - Medvin Clinical Research /ID# 205731, Whittier, California
  - Rheumatology Consultants of De /ID# 208238, Lewes, Delaware
  - Bay Area Arthritis and Osteo /ID# 208111, Brandon, Florida
  - Clinical Res of West FL, Inc. /ID# 167462, Clearwater, Florida
  - Omega Research Maitland, LLC /ID# 167376, DeBary, Florida
  - Riverside Clinical Research /ID# 167982, Edgewater, Florida
  - Lakes Research, LLC /ID# 170660, Miami, Florida
  - Kendall South Medical Center, Inc. /ID# 206857, Miami, Florida
  - Medallion Clinical Research Institute, LLC /ID# 201710, Naples, Florida
  - Rheum Assoc of Central FL /ID# 170858, Orlando, Florida
  - HMD Research LLC /ID# 208381, Orlando, Florida
  - International Medical Research - Ormond /ID# 170864, Ormond Beach, Florida
  - Millennium Research /ID# 167453, Ormond Beach, Florida
  - Arthritis Center, Inc. /ID# 170695, Palm Harbor, Florida
  - Integral Rheumatology & Immunology Specialists /ID# 206724, Plantation, Florida
  - BayCare Medical Group /ID# 170860, St. Petersburg, Florida
  - St. Anthony Comprehensive Rese /ID# 170668, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc /ID# 169099, Tampa, Florida
  - ForCare Clinical Research /ID# 206280, Tampa, Florida
  - Florida Medical Clinic /ID# 206279, Zephyrhills, Florida
  - Institute of Arthritis Researc /ID# 170694, Idaho Falls, Idaho
  - Great Lakes Clinical Trials /ID# 167471, Chicago, Illinois
  - Clinical Investigation Specialists - Skokie /ID# 167468, Skokie, Illinois
  - Deerbrook Medical Associates /ID# 207098, Vernon Hills, Illinois
  - PRN of Kansas /ID# 167985, Wichita, Kansas
  - The Arthritis & Diabetes Clinic, Inc. /ID# 170682, Monroe, Louisiana
  - Mansfield Health Center /ID# 167372, Mansfield, Massachusetts
  - Advanced Clinical Care /ID# 167367, Worcester, Massachusetts
  - June DO, PC /ID# 170670, Lansing, Michigan
  - Beals Instititute /ID# 170658, Lansing, Michigan
  - Arthritis Associates /ID# 209075, Hattiesburg, Mississippi
  - North Mississippi Med Clinics /ID# 167377, Tupelo, Mississippi
  - Clayton Medical Associates dba Saint Louis Rheumatology /ID# 170650, St Louis, Missouri
  - Physician Research Collaboration, LLC /ID# 200480, Lincoln, Nebraska
  - Dhmc /Id# 167476, Lebanon, New Hampshire
  - Ocean Rheumatology /ID# 170673, Toms River, New Jersey
  - Arthritis and Osteo Assoc /ID# 167443, Las Cruces, New Mexico
  - DJL Clinical Research, PLLC /ID# 167374, Charlotte, North Carolina
  - EmergeOrtho, P.A. /ID# 209154, Durham, North Carolina
  - Cape Fear Arthritis Care /ID# 167413, Leland, North Carolina
  - New Horizons Clinical Research /ID# 170862, Blue Ash, Ohio
  - Marietta Memorial Hospital /ID# 210968, Marietta, Ohio
  - STAT Research, Inc. /ID# 200485, Vandalia, Ohio
  - Health Research of Oklahoma /ID# 167370, Oklahoma City, Oklahoma
  - Clinical Research Ctr Reading /ID# 170708, Wyomissing, Pennsylvania
  - West Tennessee Research Inst /ID# 167366, Jackson, Tennessee
  - Nashville Arthritis and Rheumatology /ID# 206699, Nashville, Tennessee
  - Amarillo Ctr for Clin Research /ID# 200484, Amarillo, Texas
  - Tekton Research, Inc. /ID# 167475, Austin, Texas
  - Trinity Universal Res Assoc /ID# 209252, Carrollton, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 209401, College Station, Texas
  - Metroplex Clinical Research /ID# 167458, Dallas, Texas
  - Rheumatic Disease Clin Res Ctr /ID# 167474, Houston, Texas
  - Rheumatology Clinic of Houston /ID# 203689, Houston, Texas
  - Accurate Clinical Research /ID# 207059, Houston, Texas
  - West Texas Clinical Research /ID# 205732, Lubbock, Texas
  - SW Rheumatology Res. LLC /ID# 167383, Mesquite, Texas
  - Trinity Universal Research Association /ID# 209253, Plano, Texas
  - Sun Research Institute /ID# 170667, San Antonio, Texas
  - Accurate Clinical Management /ID# 200481, San Antonio, Texas
  - DM Clinical Research /ID# 167444, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 167407, Waco, Texas
  - Tidewater Physicians Medical Center /ID# 210884, Newport News, Virginia
  - Western Washington Arthritis C /ID# 205821, Bothell, Washington
  - Arthritis Northwest, PLLC /ID# 200479, Spokane, Washington
  - Rheumatology and Pulmonary cli /ID# 170863, Beckley, West Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 167385, Franklin, Wisconsin
- Belgium (4):
  - CUB Hospital Erasme /ID# 201965, Brussels, Brussels Capital
  - Cliniques Universitaires Saint Luc /ID# 201756, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Ghent /ID# 201757, Ghent, Oost-Vlaanderen
  - UZ Leuven /ID# 201927, Leuven
- Canada (6):
  - Rheumatology Research Assoc /ID# 207299, Edmonton, Alberta
  - Manitoba Clinic /ID# 202126, Winnipeg, Manitoba
  - CIADS Research Co Ltd /ID# 202125, Winnipeg, Manitoba
  - Credit Valley Rheumatology /ID# 202124, Mississauga, Ontario
  - Mount Sinai Hosp.-Toronto /ID# 202652, Toronto, Ontario
  - Dr. Latha Naik /ID# 212972, Saskatoon, Saskatchewan
- Czechia (4):
  - Revmatolog s.r.o. /ID# 202610, Jihlava, Jihlava
  - Revmatologicky ustav Praha /ID# 202142, Prague, Praha 2
  - Revmatologie MUDr. Klara Sirova /ID# 205185, Ostrava
  - CCR Czech a.s /ID# 202144, Pardubice
- Hungary (5):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 202439, Miskolc, Borsod-Abauj Zemplen county
  - Szabolcs-Szatmar-Bereg Megyei Korhazak & Egyetemi Oktatokorhaz /ID# 202441, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Revita Reumatologiai Rendelo /ID# 202438, Budapest
  - CMED Rehabilitacios es Diagnosztikai Kozpont /ID# 205804, Székesfehérvár
  - Vital Medical Center Orvosi-es Fogaszati Kozpont /ID# 202437, Veszprém
- Poland (5):
  - Malopolskie Centrum Kliniczne /ID# 206473, Krakow, Lesser Poland Voivodeship
  - McBk Sc /Id# 212575, Grodzisk Mazowiecki, Masovian Voivodeship
  - NBR Polska /ID# 206476, Warsaw, Masovian Voivodeship
  - ClinicMed Daniluk, Nowak Sp.j. /ID# 212576, Bialystok, Podlaskie Voivodeship
  - Reumatika - Centrum Reumatologii NZOZ /ID# 206472, Warsaw
- GCM Medical Group, PSC /ID# 167983, San Juan, Puerto Rico
- Spain (9):
  - Hospital Universitario A Coruña - CHUAC /ID# 202140, A Coruña, A Coruna
  - Hospital Unversitario Marques de Valdecilla /ID# 202133, Santander, Cantabria
  - Hospital Regional de Malaga /ID# 202137, Málaga, Malaga
  - Hospital Clinic /ID# 206575, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 206535, Barcelona
  - Hospital Universitario Basurto /ID# 206462, Bilbao
  - Hospital Universitario Virgen de las Nieves /ID# 209705, Granada
  - Hospital Clinico Universitario San Carlos /ID# 202135, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 202139, Valencia
- United Kingdom (3):
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 201976, Newcastle upon Tyne
  - University of Oxford /ID# 201974, Oxford
  - Warrington and Halton Teaching Hosp NHS Foundation Trust /ID# 206002, Warrington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Fleischmann R, Friedman A, Drescher E, Singhal A, Cortes-Maisonet G, Doan T, Lu W, Wang Z, Nader A, Housley W, Cohen S, Taylor PC, Blanco R. Safety and efficacy of elsubrutinib or upadacitinib alone or in combination (ABBV-599) in patients with rheumatoid arthritis and inadequate response or intolerance to biological therapies: a multicentre, double-blind, randomised, controlled, phase 2 trial. Lancet Rheumatol. 2022 Jun;4(6):e395-e406. doi: 10.1016/S2665-9913(22)00092-3. Epub 2022 Apr 27. PMID 38293957

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: all randomized participants who received at least 1 dose of randomized study drug
Period: Overall Study
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Started | 19 | 62 | 41 | 39 | 41 | 40
Completed | 17 | 58 | 38 | 34 | 35 | 38
Not Completed | 2 | 4 | 3 | 5 | 6 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 4 | 0 | 1
Not completed — Other, not specified | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least 1 dose of randomized study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo | Total
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.12) | 56.2 (12.82) | 59.2 (11.11) | 59.7 (10.95) | 58.1 (11.01) | 57.7 (10.60) | 58.0 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 48 | 36 | 35 | 33 | 35 | 204
  Male | 2 | 14 | 5 | 4 | 8 | 5 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 58 | 36 | 35 | 35 | 37 | 220
  Black or African American | 0 | 3 | 4 | 4 | 3 | 3 | 17
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Multiple | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) at Week 12
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of randomized study drug, had non-missing baseline values, and at least one post-baseline value. Baseline is defined as the last non-missing value prior to the first dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 18 | 54 | 35 | 29 | 34 | 37
units on a scale | -1.12 [-1.64 to -0.60] | -2.56 [-2.86 to -2.26] | -1.52 [-1.89 to -1.15] | -1.32 [-1.71 to -0.93] | -1.33 [-1.70 to -0.97] | -2.87 [-3.23 to -2.51]
Statistical Analysis 1: Comparison: ELS Placebo/UPA Placebo vs UPA 15 mg/ELS 60 mg; Mixed-Effect Model Repeated Measure (MMRM) analysis was conducted, testing the superiority of the combination of upadacitinib 15 mg and elsubrutinib 60 mg compared to placebo at Week 12. Data collected after a participant discontinued study drug was considered as missing. The mixed model included the categorical fixed effects of treatment, visit and treatment-by-visit interaction, prior bDMARD use, and baseline DAS28 (CRP) measurement; Test type: Superiority; p < 0.001, t-test, 2 sided; LS Mean Difference = -1.44, 90% CI 2-sided [-2.03 to -0.85], Standard Error of Mean 0.36

2. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 18 | 57 | 38 | 35 | 37 | 37
units on a scale
  Week 2: number analyzed (Participants) | 17 | 56 | 38 | 35 | 35 | 37
  Week 2 | -6.08 [-10.48 to -1.67] | -16.00 [-18.53 to -13.47] | -8.95 [-11.99 to -5.91] | -7.36 [-10.44 to -4.27] | -8.38 [-11.48 to -5.28] | -14.03 [-17.04 to -11.02]
  Week 4: number analyzed (Participants) | 17 | 57 | 37 | 34 | 37 | 37
  Week 4 | -11.60 [-16.38 to -6.82] | -20.24 [-22.97 to -17.50] | -11.67 [-15.01 to -8.34] | -10.10 [-13.50 to -6.70] | -12.90 [-16.22 to -9.58] | -20.30 [-23.57 to -17.03]
  Week 8: number analyzed (Participants) | 17 | 56 | 35 | 31 | 35 | 37
  Week 8 | -12.46 [-17.52 to -7.40] | -24.95 [-27.86 to -22.05] | -15.07 [-18.65 to -11.49] | -17.10 [-20.83 to -13.38] | -14.84 [-18.42 to -11.26] | -23.72 [-27.20 to -20.24]
  Week 12: number analyzed (Participants) | 18 | 52 | 35 | 29 | 33 | 36
  Week 12 | -14.57 [-19.77 to -9.36] | -27.00 [-30.05 to -23.95] | -17.50 [-21.22 to -13.78] | -16.70 [-20.62 to -12.78] | -16.51 [-20.27 to -12.75] | -28.85 [-32.48 to -25.21]

3. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: The SDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global disease activity assessed by the participant on a visual analogue scale from 0 to 10 (cm), global disease activity assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein (CRP; mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86.with higher scores indicating higher disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 18 | 57 | 38 | 35 | 37 | 37
units on a scale
  Week 2: number analyzed (Participants) | 17 | 56 | 38 | 35 | 35 | 37
  Week 2 | -6.17 [-10.67 to -1.67] | -17.01 [-19.60 to -14.43] | -8.79 [-11.89 to -5.68] | -7.42 [-10.57 to -4.26] | -8.54 [-11.71 to -5.38] | -15.30 [-18.37 to -12.22]
  Week 4: number analyzed (Participants) | 17 | 57 | 37 | 34 | 37 | 37
  Week 4 | -11.80 [-16.67 to -6.93] | -21.24 [-24.02 to -18.45] | -11.46 [-14.85 to -8.06] | -10.15 [-13.61 to -6.68] | -12.87 [-16.25 to -9.49] | -21.59 [-24.92 to -18.26]
  Week 8: number analyzed (Participants) | 17 | 56 | 35 | 30 | 35 | 37
  Week 8 | -12.15 [-17.35 to -6.95] | -25.96 [-28.95 to -22.98] | -15.26 [-18.94 to -11.57] | -17.32 [-21.17 to -13.46] | -15.21 [-18.89 to -11.53] | -25.07 [-28.65 to -21.49]
  Week 12: number analyzed (Participants) | 18 | 52 | 35 | 29 | 32 | 36
  Week 12 | -14.44 [-19.84 to -9.04] | -28.06 [-31.22 to -24.89] | -18.01 [-21.86 to -14.15] | -17.12 [-21.20 to -13.05] | -16.73 [-20.65 to -12.81] | -29.65 [-33.42 to -25.88]

4. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) at Week 12
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Clinical remission (CR) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than 2.6.
Time Frame: At Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of randomized study drug, nonresponder imputation was used for missing data
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants | 10.5 [3.55 to 27.35] | 32.3 [23.41 to 42.59] | 19.5 [11.36 to 31.44] | 7.7 [3.12 to 17.76] | 9.8 [4.46 to 20.04] | 42.5 [30.52 to 55.43]

5. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Disease Activity Score 28 C-reactive Protein [DAS28-CRP]) at Week 12
Description: The DAS28-CRP is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Scores on the DAS28-CRP range from 0 to approximately 10, where higher scores indicate more disease activity. Low Disease Activity (LDA) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than or equal to 3.2.
Time Frame: At Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants | 21.1 [9.82 to 39.50] | 41.9 [32.18 to 52.37] | 22.0 [13.24 to 34.13] | 10.3 [4.69 to 20.98] | 14.6 [7.76 to 25.89] | 55.0 [42.16 to 67.21]

6. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on Clinical Disease Activity Index (CDAI) Criteria
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. Low Disease Activity (LDA) based on CDAI is defined as achieving a CDAI of less than or equal to 10.
Time Frame: Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 10.5 [3.55 to 27.35] | 16.1 [9.89 to 25.20] | 9.8 [4.46 to 20.04] | 0 [0.00 to 6.49] | 2.4 [0.55 to 10.22] | 12.5 [6.22 to 23.53]
  Week 4 | 10.5 [3.55 to 27.35] | 29.0 [20.59 to 39.23] | 12.2 [6.06 to 23.01] | 7.7 [3.12 to 17.76] | 12.2 [6.06 to 23.01] | 22.5 [13.59 to 34.90]
  Week 8 | 5.3 [1.18 to 20.50] | 46.8 [36.71 to 57.11] | 17.1 [9.53 to 28.69] | 20.5 [11.96 to 32.89] | 24.4 [15.17 to 36.78] | 35.0 [23.91 to 47.99]
  Week 12 | 26.3 [13.44 to 45.09] | 37.1 [27.74 to 47.53] | 34.1 [23.29 to 46.97] | 17.9 [10.03 to 30.02] | 17.1 [9.53 to 28.69] | 57.5 [44.57 to 69.48]

7. Secondary Outcome: Percentage of Participants Achieving Complete Remission (CR) Based on Clinical Disease Activity Index (CDAI) Criteria
Description: The CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. Complete Remission (CR) based on CDAI is defined as achieving a CDAI of less than or equal to 2.8.
Time Frame: Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 0 [0.00 to 12.46] | 3.2 [1.07 to 9.29] | 0 [0.00 to 6.19] | 0 [0.00 to 6.49] | 0 [0.00 to 6.19] | 0 [0.00 to 6.34]
  Week 4 | 0 [0.00 to 12.46] | 6.5 [2.93 to 13.62] | 2.4 [0.55 to 10.22] | 2.6 [0.57 to 10.71] | 0 [0.00 to 6.19] | 2.5 [0.56 to 10.46]
  Week 8 | 0 [0.00 to 12.46] | 12.9 [7.43 to 21.48] | 7.3 [2.96 to 16.96] | 2.6 [0.57 to 10.71] | 2.4 [0.55 to 10.22] | 12.5 [6.22 to 23.53]
  Week 12 | 5.3 [1.18 to 20.50] | 14.5 [8.65 to 23.35] | 7.3 [2.96 to 16.96] | 5.1 [1.71 to 14.37] | 0 [0.00 to 6.19] | 15.0 [7.96 to 26.47]

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the American College of Rheumatology 20% response (ACR20) criteria:
  1. ≥ 20% improvement in 68-tender joint count
  2. ≥ 20% improvement in 66-swollen joint count and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 21.1 [9.82 to 39.50] | 45.2 [35.19 to 55.54] | 24.4 [15.17 to 36.78] | 12.8 [6.38 to 24.08] | 14.6 [7.76 to 25.89] | 52.5 [39.77 to 64.91]
  Week 4 | 42.1 [25.63 to 60.55] | 51.6 [41.33 to 61.76] | 29.3 [19.16 to 41.94] | 23.1 [13.95 to 35.70] | 22.0 [13.24 to 34.13] | 55.0 [42.16 to 67.21]
  Week 8 | 36.8 [21.37 to 55.59] | 64.5 [54.11 to 73.71] | 39.0 [27.55 to 51.86] | 30.8 [20.20 to 43.84] | 39.0 [27.55 to 51.86] | 67.5 [54.55 to 78.23]
  Week 12 | 47.4 [30.07 to 65.33] | 64.5 [54.11 to 73.71] | 41.5 [29.72 to 54.26] | 30.8 [20.20 to 43.84] | 34.1 [23.29 to 46.97] | 72.5 [59.75 to 82.40]

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the American College of Rheumatology 50% response (ACR50) criteria:
  1. ≥ 50% improvement in 68-tender joint count
  2. ≥ 50% improvement in 66-swollen joint count and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 0 [0.00 to 12.46] | 16.1 [9.89 to 25.20] | 4.9 [1.63 to 13.71] | 0 [0.00 to 6.49] | 0 [0.00 to 6.19] | 12.5 [6.22 to 23.53]
  Week 4 | 10.5 [3.55 to 27.35] | 19.4 [12.46 to 28.82] | 17.1 [9.53 to 28.69] | 2.6 [0.57 to 10.71] | 4.9 [1.63 to 13.71] | 30.0 [19.66 to 42.87]
  Week 8 | 5.3 [1.18 to 20.50] | 41.9 [32.18 to 52.37] | 19.5 [11.36 to 31.44] | 12.8 [6.38 to 24.08] | 7.3 [2.96 to 16.96] | 40.0 [28.29 to 52.98]
  Week 12 | 21.1 [9.82 to 39.50] | 45.2 [35.19 to 55.54] | 29.3 [19.16 to 41.94] | 12.8 [6.38 to 24.08] | 17.1 [9.53 to 28.69] | 47.5 [35.09 to 60.23]

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the American College of Rheumatology 70% response (ACR70) criteria:
  1. ≥ 70% improvement in 68-tender joint count
  2. ≥ 70% improvement in 66-swollen joint count and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Patient's Assessment of Pain (Visual Analog Scale [VAS])
     * Patient's Global Assessment of Disease Activity (PtGA)
     * Physician's Global Assessment of Disease Activity (PhGA)
     * Health Assessment Questionnaire Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP)
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 0 [0.00 to 12.46] | 8.1 [3.98 to 15.66] | 2.4 [0.55 to 10.22] | 0 [0.00 to 6.49] | 0 [0.00 to 6.19] | 0 [0.00 to 6.34]
  Week 4 | 0 [0.00 to 12.46] | 9.7 [5.09 to 17.64] | 4.9 [1.63 to 13.71] | 2.6 [0.57 to 10.71] | 0 [0.00 to 6.19] | 15.0 [7.96 to 26.47]
  Week 8 | 0 [0.00 to 12.46] | 17.7 [11.16 to 27.02] | 4.9 [1.63 to 13.71] | 2.6 [0.57 to 10.71] | 0 [0.00 to 6.19] | 25.0 [15.57 to 37.60]
  Week 12 | 15.8 [6.49 to 33.62] | 25.8 [17.81 to 35.82] | 14.6 [7.76 to 25.89] | 5.1 [1.71 to 14.37] | 9.8 [4.46 to 20.04] | 27.5 [17.60 to 40.25]

11. Secondary Outcome: Change From Baseline in Tender Joint Count 68 (TJC68)
Description: Sixty-eight joints were assessed for tenderness by physical examination. Pain or tenderness of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with tenderness) to 68 (worst possible score/68 joints with tenderness). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: tender joint counts
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 61 | 39 | 37 | 40 | 40
tender joint counts
  Week 2: number analyzed (Participants) | 19 | 61 | 39 | 37 | 39 | 40
  Week 2 | -2.47 [-6.10 to 1.16] | -8.42 [-10.53 to -6.31] | -3.65 [-6.23 to -1.07] | -3.86 [-6.46 to -1.26] | -4.88 [-7.43 to -2.33] | -8.57 [-11.09 to -6.05]
  Week 4: number analyzed (Participants) | 19 | 61 | 38 | 36 | 40 | 39
  Week 4 | -9.21 [-13.08 to -5.34] | -11.86 [-14.10 to -9.62] | -5.16 [-7.93 to -2.39] | -5.39 [-8.18 to -2.60] | -8.08 [-10.77 to -5.39] | -12.76 [-15.46 to -10.06]
  Week 8: number analyzed (Participants) | 18 | 59 | 36 | 33 | 38 | 38
  Week 8 | -8.82 [-12.85 to -4.79] | -15.44 [-17.75 to -13.12] | -8.43 [-11.31 to -5.55] | -10.83 [-13.78 to -7.88] | -9.08 [-11.88 to -6.27] | -14.76 [-17.56 to -11.97]
  Week 12: number analyzed (Participants) | 18 | 56 | 36 | 31 | 35 | 37
  Week 12 | -8.47 [-12.81 to -4.12] | -16.33 [-18.84 to -13.83] | -9.14 [-12.23 to -6.05] | -9.33 [-12.55 to -6.12] | -12.58 [-15.64 to -9.52] | -17.56 [-20.58 to -14.53]

12. Secondary Outcome: Change From Baseline in Swollen Joint Count 66 (SJC66)
Description: Sixty-six joints were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with swelling) to 66 (worst possible score/66 joints with swelling). Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: swollen joint counts
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 61 | 39 | 37 | 40 | 40
swollen joint counts
  Week 2: number analyzed (Participants) | 19 | 61 | 39 | 37 | 39 | 40
  Week 2 | -3.12 [-5.20 to -1.05] | -6.06 [-7.26 to -4.86] | -3.61 [-5.08 to -2.14] | -3.30 [-4.78 to -1.82] | -4.13 [-5.60 to -2.67] | -6.02 [-7.46 to -4.58]
  Week 4: number analyzed (Participants) | 19 | 61 | 38 | 36 | 40 | 39
  Week 4 | -4.70 [-6.92 to -2.49] | -7.96 [-9.24 to -6.68] | -5.11 [-6.69 to -3.53] | -4.67 [-6.27 to -3.07] | -6.05 [-7.60 to -4.51] | -8.81 [-10.35 to -7.26]
  Week 8: number analyzed (Participants) | 18 | 59 | 36 | 33 | 38 | 38
  Week 8 | -4.32 [-6.57 to -2.06] | -10.28 [-11.57 to -8.99] | -6.15 [-7.77 to -4.54] | -8.08 [-9.74 to -6.42] | -7.58 [-9.15 to -6.00] | -10.11 [-11.68 to -8.55]
  Week 12: number analyzed (Participants) | 18 | 56 | 36 | 31 | 35 | 37
  Week 12 | -5.58 [-8.05 to -3.11] | -10.86 [-12.29 to -9.44] | -6.68 [-8.44 to -4.92] | -7.85 [-9.70 to -6.01] | -8.59 [-10.35 to -6.83] | -11.14 [-12.86 to -9.42]

13. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain (Visual Analog Scale [VAS])
Description: Participants rated their pain on a visual analogue scale (VAS) of 0 to 100 (mm), with 0 representing no pain and 100 representing the worst possible pain. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 35 | 40 | 39
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 35 | 38 | 39
  Week 2 | -14.97 [-22.80 to -7.14] | -24.02 [-28.63 to -19.41] | -10.22 [-15.81 to -4.63] | -8.78 [-14.49 to -3.07] | -7.61 [-13.12 to -2.11] | -15.99 [-21.49 to -10.48]
  Week 4: number analyzed (Participants) | 19 | 59 | 37 | 34 | 40 | 39
  Week 4 | -20.87 [-29.60 to -12.14] | -28.17 [-33.28 to -23.07] | -12.95 [-19.27 to -6.63] | -8.41 [-14.85 to -1.97] | -9.91 [-15.93 to -3.88] | -25.58 [-31.69 to -19.48]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 31 | 38 | 38
  Week 8 | -16.21 [-25.97 to -6.45] | -31.86 [-37.50 to -26.22] | -20.92 [-27.96 to -13.88] | -11.12 [-18.46 to -3.79] | -13.90 [-20.64 to -7.16] | -30.70 [-37.47 to -23.92]
  Week 12: number analyzed (Participants) | 18 | 54 | 35 | 29 | 35 | 37
  Week 12 | -23.37 [-33.74 to -13.01] | -32.27 [-38.32 to -26.23] | -19.52 [-26.97 to -12.06] | -10.46 [-18.38 to -2.55] | -17.84 [-25.13 to -10.55] | -38.34 [-45.57 to -31.12]

14. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity (PGA)
Description: Participants rated their disease activity for the past 24 hours using a Patient's Global Assessment of Disease Activity Global visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 35 | 40 | 39
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 35 | 38 | 39
  Week 2 | -11.87 [-20.12 to -3.63] | -23.44 [-28.31 to -18.57] | -11.16 [-17.07 to -5.25] | -6.47 [-12.51 to -0.44] | -5.95 [-11.76 to -0.14] | -14.76 [-20.56 to -8.95]
  Week 4: number analyzed (Participants) | 19 | 59 | 37 | 34 | 40 | 39
  Week 4 | -20.93 [-29.91 to -11.94] | -25.97 [-31.24 to -20.70] | -12.79 [-19.32 to -6.26] | -7.15 [-13.79 to -0.50] | -8.73 [-14.94 to -2.51] | -23.02 [-29.31 to -16.73]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 31 | 38 | 38
  Week 8 | -15.14 [-25.37 to -4.91] | -28.05 [-33.97 to -22.13] | -17.25 [-24.65 to -9.84] | -6.27 [-14.00 to 1.45] | -14.25 [-21.34 to -7.17] | -26.79 [-33.90 to -19.69]
  Week 12: number analyzed (Participants) | 18 | 54 | 35 | 29 | 35 | 37
  Week 12 | -19.55 [-30.15 to -8.95] | -30.52 [-36.72 to -24.32] | -19.47 [-27.13 to -11.81] | -8.45 [-16.58 to -0.33] | -16.40 [-23.89 to -8.92] | -33.53 [-40.94 to -26.13]

15. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity (PhGA)
Description: The physician assessed a participant's disease activity at the time of the visit using a Physician's Global Assessment of Disease visual analogue scale (VAS). The range is 0 to 100 mm, with 0 representing no disease activity and 100 representing severe disease activity. Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 18 | 58 | 38 | 35 | 37 | 38
units on a scale
  Week 2: number analyzed (Participants) | 17 | 57 | 38 | 35 | 36 | 38
  Week 2 | -16.31 [-24.67 to -7.96] | -22.35 [-27.10 to -17.60] | -19.01 [-24.74 to -13.27] | -16.12 [-21.97 to -10.26] | -11.64 [-17.44 to -5.84] | -24.71 [-30.37 to -19.05]
  Week 4: number analyzed (Participants) | 17 | 58 | 37 | 34 | 37 | 37
  Week 4 | -25.20 [-33.52 to -16.89] | -33.54 [-38.26 to -28.82] | -25.33 [-31.11 to -19.55] | -19.59 [-25.49 to -13.69] | -18.31 [-24.05 to -12.56] | -34.17 [-39.86 to -28.49]
  Week 8: number analyzed (Participants) | 17 | 57 | 35 | 31 | 35 | 37
  Week 8 | -24.47 [-32.71 to -16.22] | -40.00 [-44.71 to -35.29] | -30.06 [-35.91 to -24.22] | -33.93 [-39.99 to -27.87] | -25.21 [-31.03 to -19.40] | -41.02 [-46.69 to -35.36]
  Week 12: number analyzed (Participants) | 18 | 53 | 35 | 29 | 33 | 36
  Week 12 | -23.19 [-31.69 to -14.69] | -46.98 [-52.00 to -41.96] | -30.15 [-36.28 to -24.03] | -31.68 [-38.19 to -25.18] | -24.55 [-30.75 to -18.36] | -50.89 [-56.87 to -44.91]

16. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from baseline in the overall score indicates improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 35 | 40 | 38
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 35 | 38 | 38
  Week 2 | -0.22 [-0.37 to -0.06] | -0.34 [-0.43 to -0.25] | -0.13 [-0.24 to -0.02] | -0.06 [-0.17 to 0.05] | -0.16 [-0.27 to -0.05] | -0.22 [-0.33 to -0.11]
  Week 4: number analyzed (Participants) | 19 | 59 | 37 | 34 | 40 | 38
  Week 4 | -0.36 [-0.53 to -0.18] | -0.39 [-0.49 to -0.29] | -0.11 [-0.23 to 0.02] | -0.14 [-0.27 to -0.02] | -0.21 [-0.33 to -0.09] | -0.33 [-0.45 to -0.20]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 31 | 38 | 37
  Week 8 | -0.24 [-0.44 to -0.05] | -0.47 [-0.59 to -0.36] | -0.29 [-0.43 to -0.15] | -0.15 [-0.30 to -0.00] | -0.15 [-0.29 to -0.02] | -0.47 [-0.61 to -0.33]
  Week 12: number analyzed (Participants) | 18 | 54 | 35 | 29 | 35 | 36
  Week 12 | -0.30 [-0.52 to -0.08] | -0.52 [-0.65 to -0.39] | -0.31 [-0.46 to -0.15] | -0.12 [-0.28 to 0.05] | -0.18 [-0.33 to -0.03] | -0.54 [-0.70 to -0.39]

17. Secondary Outcome: Change From Baseline in High-Sensitivity C-reactive Protein (hsCRP)
Description: C-reactive protein is a blood test marker for inflammation in the body, and levels rise in response to inflammation. A negative change from baseline in indicates improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/L
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 61 | 39 | 37 | 40 | 40
mg/L
  Week 2: number analyzed (Participants) | 19 | 61 | 39 | 37 | 39 | 40
  Week 2 | -0.51 [-4.82 to 3.81] | -9.29 [-11.79 to -6.80] | 2.26 [-0.81 to 5.33] | -0.34 [-3.43 to 2.74] | -0.72 [-3.74 to 2.30] | -12.27 [-15.26 to -9.27]
  Week 4: number analyzed (Participants) | 19 | 61 | 38 | 36 | 40 | 39
  Week 4 | 1.54 [-3.72 to 6.79] | -10.08 [-13.08 to -7.08] | 2.71 [-1.05 to 6.46] | -0.78 [-4.58 to 3.02] | 0.72 [-2.91 to 4.35] | -12.59 [-16.27 to -8.92]
  Week 8: number analyzed (Participants) | 18 | 59 | 36 | 32 | 38 | 38
  Week 8 | 3.23 [-1.56 to 8.03] | -9.97 [-12.70 to -7.24] | -1.39 [-4.83 to 2.05] | -2.58 [-6.15 to 1.00] | -2.93 [-6.26 to 0.39] | -13.13 [-16.46 to -9.81]
  Week 12: number analyzed (Participants) | 18 | 56 | 36 | 31 | 34 | 37
  Week 12 | 1.45 [-5.10 to 8.00] | -10.95 [-14.73 to -7.18] | -4.58 [-9.26 to 0.09] | -5.78 [-10.77 to -0.78] | -0.81 [-5.58 to 3.97] | -7.44 [-12.03 to -2.86]

18. Secondary Outcome: Change From Baseline in Disease Activity Score 28 C-reactive Protein [DAS28-CRP])
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 35 | 40 | 39
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 35 | 38 | 39
  Week 2 | -0.46 [-0.83 to -0.10] | -1.53 [-1.75 to -1.31] | -0.63 [-0.89 to -0.36] | -0.44 [-0.71 to -0.18] | -0.56 [-0.82 to -0.30] | -1.43 [-1.69 to -1.17]
  Week 4: number analyzed (Participants) | 19 | 59 | 37 | 34 | 40 | 39
  Week 4 | -0.90 [-1.33 to -0.47] | -1.96 [-2.21 to -1.71] | -0.87 [-1.18 to -0.56] | -0.68 [-1.00 to -0.36] | -0.82 [-1.11 to -0.52] | -1.98 [-2.28 to -1.67]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 30 | 38 | 38
  Week 8 | -0.78 [-1.27 to -0.29] | -2.40 [-2.68 to -2.11] | -1.21 [-1.56 to -0.86] | -1.24 [-1.61 to -0.87] | -1.11 [-1.45 to -0.77] | -2.34 [-2.68 to -2.00]
  Week 12: number analyzed (Participants) | 18 | 54 | 35 | 29 | 34 | 37
  Week 12 | -1.12 [-1.64 to -0.60] | -2.56 [-2.86 to -2.26] | -1.52 [-1.89 to -1.15] | -1.32 [-1.71 to -0.93] | -1.33 [-1.70 to -0.97] | -2.87 [-3.23 to -2.51]

19. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Erythrocyte Sedimentation Rate (DAS28- ESR)
Description: The DAS28-ESR is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR; mm/hour), and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 100 mm) are included in the DAS28 -ESR score. Scores on the DAS28-ESR range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 34 | 40 | 39
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 34 | 38 | 39
  Week 2 | -0.46 [-0.82 to -0.09] | -1.48 [-1.69 to -1.26] | -0.52 [-0.79 to -0.26] | -0.46 [-0.74 to -0.19] | -0.57 [-0.83 to -0.32] | -1.32 [-1.58 to -1.06]
  Week 4: number analyzed (Participants) | 19 | 58 | 37 | 34 | 40 | 39
  Week 4 | -0.86 [-1.30 to -0.43] | -1.93 [-2.19 to -1.68] | -0.79 [-1.11 to -0.48] | -0.59 [-0.91 to -0.26] | -0.92 [-1.23 to -0.62] | -1.90 [-2.20 to -1.59]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 30 | 37 | 38
  Week 8 | -0.80 [-1.29 to -0.31] | -2.41 [-2.69 to -2.12] | -1.07 [-1.42 to -0.71] | -1.15 [-1.52 to -0.78] | -1.20 [-1.54 to -0.86] | -2.31 [-2.65 to -1.97]
  Week 12: number analyzed (Participants) | 18 | 54 | 35 | 29 | 35 | 37
  Week 12 | -1.18 [-1.71 to -0.64] | -2.53 [-2.84 to -2.22] | -1.41 [-1.80 to -1.03] | -1.24 [-1.65 to -0.83] | -1.44 [-1.82 to -1.06] | -2.88 [-3.25 to -2.50]

20. Secondary Outcome: Change From Baseline in Morning Stiffness Severity
Description: Morning stiffness severity was assessed by a numeric rating-scale (NRS). Participants rated the severity of morning stiffness during the past week from 0 to 10 with 0 representing "not severe" and 10 "very severe". Negative values indicate improvement from baseline.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 59 | 39 | 35 | 40 | 38
units on a scale
  Week 2: number analyzed (Participants) | 19 | 59 | 39 | 35 | 38 | 38
  Week 2 | -1.76 [-2.54 to -0.98] | -2.02 [-2.48 to -1.56] | -0.91 [-1.47 to -0.35] | -0.68 [-1.26 to -0.11] | -0.59 [-1.15 to -0.04] | -1.84 [-2.40 to -1.29]
  Week 4: number analyzed (Participants) | 19 | 59 | 37 | 34 | 40 | 38
  Week 4 | -1.76 [-2.63 to -0.90] | -2.71 [-3.22 to -2.21] | -0.82 [-1.45 to -0.20] | -0.83 [-1.47 to -0.19] | -1.08 [-1.67 to -0.48] | -2.51 [-3.13 to -1.90]
  Week 8: number analyzed (Participants) | 18 | 57 | 35 | 31 | 38 | 37
  Week 8 | -1.67 [-2.56 to -0.77] | -3.07 [-3.59 to -2.55] | -1.30 [-1.94 to -0.65] | -0.97 [-1.64 to -0.30] | -1.50 [-2.11 to -0.88] | -3.07 [-3.70 to -2.44]
  Week 12: number analyzed (Participants) | 18 | 54 | 34 | 29 | 35 | 36
  Week 12 | -1.61 [-2.60 to -0.63] | -3.23 [-3.81 to -2.65] | -1.27 [-1.99 to -0.56] | -1.30 [-2.06 to -0.55] | -1.66 [-2.36 to -0.97] | -3.36 [-4.06 to -2.67]

21. Secondary Outcome: Percentage of Participants Achieving Minimal Clinically Important Difference (MCID) in Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. The minimal clinically important difference (MCID) in HAQ-DI is defined as change from Baseline ≤ -0.22 for rheumatoid arthritis.
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 52.6 [34.67 to 69.93] | 51.6 [41.33 to 61.76] | 36.6 [25.40 to 49.43] | 30.8 [20.20 to 43.84] | 36.6 [25.40 to 49.43] | 52.5 [39.77 to 64.91]
  Week 4 | 68.4 [49.55 to 82.70] | 54.8 [44.46 to 64.81] | 34.1 [23.29 to 46.97] | 41.0 [29.07 to 54.15] | 53.7 [41.02 to 65.84] | 45.0 [32.79 to 57.84]
  Week 8 | 52.6 [34.67 to 69.93] | 58.1 [47.63 to 67.82] | 51.2 [38.71 to 63.58] | 51.3 [38.47 to 63.93] | 36.6 [25.40 to 49.43] | 65.0 [52.01 to 76.09]
  Week 12 | 47.4 [30.07 to 65.33] | 58.1 [47.63 to 67.82] | 53.7 [41.02 to 65.84] | 43.6 [31.37 to 56.64] | 43.9 [31.93 to 56.63] | 55.0 [42.16 to 67.21]

22. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology/European League Against Rheumatism (EULAR) Boolean Remission
Description: The EULAR Boolean-based definition of remission is as follows: at any time point, a participant must satisfy all of the following: tender joint count ≤1, swollen joint count ≤1, C-reactive protein ≤1 mg/dl and Patient Global Assessment (PGA) ≤1 (on a 0-10 scale).
Time Frame: Baseline, Week 2, Week 4, Week 8, and Week 12
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
Number analyzed (Participants) | 19 | 62 | 41 | 39 | 41 | 40
percentage of participants
  Week 2 | 0 [0.00 to 12.46] | 1.6 [0.36 to 6.91] | 0 [0.00 to 6.19] | 0 [0.00 to 6.49] | 0 [0.00 to 6.19] | 0 [0.00 to 6.34]
  Week 4 | 0 [0.00 to 12.46] | 6.5 [2.93 to 13.62] | 2.4 [0.55 to 10.22] | 0 [0.00 to 6.49] | 0 [0.00 to 6.19] | 2.5 [0.56 to 10.46]
  Week 8 | 0 [0.00 to 12.46] | 6.5 [2.93 to 13.62] | 2.4 [0.55 to 10.22] | 5.1 [1.71 to 14.37] | 0 [0.00 to 6.19] | 12.5 [6.22 to 23.53]
  Week 12 | 0 [0.00 to 12.46] | 11.3 [6.24 to 19.58] | 9.8 [4.46 to 20.04] | 2.6 [0.57 to 10.71] | 2.4 [0.55 to 10.22] | 10.0 [4.57 to 20.50]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after last study drug administration, up to 16 weeks. In addition, serious adverse events and protocol-related nonserious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 30 days have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ELS Placebo/UPA Placebo | UPA 15 mg/ELS 60 mg | ELS 60 mg/UPA Placebo | ELS 20 mg/UPA Placebo | ELS 5 mg/UPA Placebo | UPA 15 mg/ELS Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/62 | 0/41 | 0/39 | 1/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/62 | 0/41 | 2/39 | 3/41 | 0/40
Other Adverse Events (participants affected / at risk) | 10/19 | 7/62 | 17/41 | 10/39 | 8/41 | 9/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELS Placebo/UPA Placebo (N=19) | UPA 15 mg/ELS 60 mg (N=62) | ELS 60 mg/UPA Placebo (N=41) | ELS 20 mg/UPA Placebo (N=39) | ELS 5 mg/UPA Placebo (N=41) | UPA 15 mg/ELS Placebo (N=40)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELS Placebo/UPA Placebo (N=19) | UPA 15 mg/ELS 60 mg (N=62) | ELS 60 mg/UPA Placebo (N=41) | ELS 20 mg/UPA Placebo (N=39) | ELS 5 mg/UPA Placebo (N=41) | UPA 15 mg/ELS Placebo (N=40)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 2 (2) | 3 (4)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BONE DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03682705/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03682705/SAP_001.pdf